CLINICAL TRIAL: NCT01329562
Title: Evaluation of CGRP, Estrogen, Cortisol, VIP, α-Amylase, PGE2, PGI2 and ß-Endorphin Levels in Saliva of Menstrual Migraine Patients Before and After Treatment With Treximet™
Brief Title: CGRP, Estrogen, Cortisol, VIP, α-Amylase, PGE2, PGI2 and ß-Endorphin Levels in Menstrual Migraine Before and After Treximet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114680
Record Dates: First submitted 2011-03-17; First posted 2011-04-06 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Menstrual Migraine
Keywords: Menstrual migraine; Menstrually-related migraine; Treximet; CGRP; calcitonin gene-related peptide
MeSH Terms: interventions — sumatriptan-naproxen; Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treximet (Active Comparator): Subjects randomized to Group A will be provided with 1 tablet of Treximet to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Interventions: Drug: Treximet
- Placebo (Placebo Comparator): Subjects randomized to Group B will be provided with 1 tablet of placebo to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treximet — Tablet for oral administration contains sumatriptan 85mg / naproxen sodium 500mg.
  Other Names: Sumatriptan/Naproxen Sodium
  Arms: Treximet
Drug: Placebo — A placebo tablet matching Treximet for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to (1) evaluate pain-free efficacy of Treximet™ following treatment of menstrual migraine, (2) investigate levels of Calcitonin gene-related peptide (CGRP), estrogen, cortisol, vasoactive intestinal peptide (VIP), alpha (a)-amylase, Prostaglandin E2 (PGE2), Prostaglandin I2 (PGI2) and beta (ß)-endorphin in saliva before and after Treximet™, (3) evaluate efficacy of Treximet™ to return to baseline levels following treatment, and (4) correlate estrogen in saliva vs. urinary estradiol at mid-luteal, onset of menstrually-related migraine, and after successful treatment with Treximet™.

DETAILED DESCRIPTION:
This double-blind multi-site study will be conducted to enroll 40 evaluable participants. All subjects will be medically stable at enrollment and be on a stabilized dosage of daily medications.

At Visit 1 (Baseline) following Informed Consent, a physical and neurological exam, baseline electrocardiogram (ECG), and vital signs will be completed. A urine pregnancy test will be collected by all subjects of childbearing potential. Routine labs (electrolyte panel with creatinine, alanine aminotransferase (ALT) / aspartate aminotransferase (AST), a luteinizing hormone (LH) lab (for menstrual cycle staging) and a baseline saliva sample (for CGRP, estrogen, cortisol, VIP, a-amylase, PGI2, PGE2 and β-endorphin analysis) will be collected. Subjects should be headache-free at Visit 1. A medical, headache, and medication history will be collected on all subjects and eligible subjects will be randomized 1:1 to Group A or Group B. Group A will receive Treximet™ (sumatriptan succinate 85 milligrams (mg) and naproxen sodium 500 mg) 1 tablet. Group B will be provided 1 matching placebo tablet. Subjects will be instructed to not start study medication until notified by study staff that lab results were normal and they are eligible to proceed. Subjects will be instructed to treat as early as possible following the onset of a typical menstrual headache. Groups A and B will be provided with Treximet™ 1 tablet for rescue between 2 and 24 hours for persistent or recurring headache. Subjects will receive a Diary and instructions on Digital Versatile Disc (DVD) regarding documentation. Migraine associated symptoms (ie nausea, vomiting, light sensitivity, or sound sensitivity) will be collected as well as sleeplessness, difficulty thinking other bodily pain, and menstrual associated symptoms (to include intensity of menstrual cramps).

Subjects will be given kits with written instructions for collection of urine and saliva samples and additional saliva instructions on DVD. All subjects will be given LH testing kits to define the time of ovulation. Diary documentation begins at the time of ovulation. They will collect baseline saliva and first morning urine samples during the mid-luteal time period for two consecutive days, which is defined as 4-7 days after the LH surge. Subjects will also be instructed to begin collection of saliva 48 hours prior to the start of menses at 8:00 am, 2:00 pm, and 8:00 pm for two days or until menstrual migraine occurs. They also will collect a first morning urine sample on the two mornings prior to menses. At the point of headache onset, subjects will be instructed to collect saliva at onset of pain, time of treatment, 2 and 24 hours following treatment, at pain free, 2 hours after pain free, and 24 hours after pain free. Subjects will also be instructed to collect a urine specimen when they are pain free following treatment with study medication. Subjects will document migraine associated symptoms, menstrual associated symptoms, and recurrence symptoms at all saliva collection time points in the provided Diary per instruction.

Subjects should be instructed to phone the study coordinator at the end of the menstrual cycle to return for Visit 2 within 7 days.

_________________________

At Visit 2 (Review) Diaries will be reviewed and frozen saliva and urine samples will be returned to the clinic. Subjects must meet the following criteria for urine and saliva analysis:

* Diary review indicates that headache would have, if left untreated, at least one symptom of migraine (nausea, vomiting, phonophobia, or photophobia) . And
* Headache was associated with the onset of menses

And

• Saliva and urine samples are returned to the clinic.

Medical and medication history will be updated and adverse events collected. A urine pregnancy test will be collected by all subjects of childbearing potential. Drug accountability and compliance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subject

1. is female between the ages of 18-45 and, if of child-bearing potential, has a negative pregnancy test (urine or serum) at screen, and agrees to one of the following:

   * Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study,
   * History of bilateral tubal ligation
   * Sterilization of male partner; or,
   * Implants of levonorgestrel; or,
   * Injectable progestogen; or,
   * Oral contraceptive (combination therapy with ethinyl estradiol plus a progestin) with a placebo week every 1-3 months; or,
   * Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or,
   * Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm); or,
   * Any other barrier methods (only if used in combination with any of the above acceptable methods); or,
   * Any other methods with published data showing that the highest expected failure rate for that method is less than 1% per year.
2. is formally diagnosed with International Classification of Headache Disorders (ICHD) menstrual migraine
3. has regular and predictable monthly menstrual cycles within a range of 22-32 days for the past 3 cycles.
4. has fewer than 15 headache days per month in past 3 months
5. has headache that, if left untreated, would have at least 1 symptom of migraine (nausea, vomiting, photophobia, or phonophobia) or respond to a triptan or ergotamine-containing medication with at least 50% of headaches
6. has a history of reliably predicting menstrual migraine headache onset at least 70% of the time
7. is medically stable as determined by the Investigator
8. if taking any concomitant medications, is on a stabilized dosage at the discretion of the investigator
9. is able to understand and communicate intelligibly with the study observer
10. is able to take oral medication, adhere to the medication regimens and perform study procedures
11. is able to read and comprehend written instructions and be willing to complete all procedures and assessments required by this protocol
12. is able to demonstrate the willingness to participate by signing and understanding an informed consent after full explanation of the study

Exclusion Criteria:

Subject

1. has a history of serotonin syndrome.
2. has any medical condition that, in the opinion of the investigator, could alter the response to study medication or confound the results of the study (ie. pathology of the salivary glands such as viral or bacterial sialadenitis or obstructive sialadenitis or Sjögren's Syndrome)
3. is of childbearing potential and not using adequate contraceptive measures
4. has history of retinal, basilar or hemiplegic migraine, cluster headache, or secondary headaches (such as due to trauma, infection, alterations of homeostasis, ear, nose and throat (ENT) or psychiatric disorders, cranial or cervical disorders or neuralgias)
5. in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or the presence of risk factors including but not limited to, hypertension, hypercholesterolemia, smoker, obesity, diabetes, or family history of coronary artery disease)
6. has blood pressure equal to or greater than 160/90 millimeters of mercury (mmHg) in 2 out of 3 blood pressure (BP) measurements at screening or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker
7. has a history of significant congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study
8. has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with any of the above
9. has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold; or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening
10. has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study
11. has hypersensitivity, intolerance, or contraindication to the use of any triptan, non-steroidal anti-inflammatory drug (NSAID) or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma
12. is currently taking, or has taken in the previous three months, a migraine prophylactic medication containing methysergide; or is taking a migraine or menstrual migraine prophylactic medication that is not stabilized (eg. Perimenstrual use of triptans and estradiol patches)
13. has a recent history of regular use of opioids or barbiturates for treatment of their migraine headache and/or other non-migraine pain or any medication overuse that in the opinion of the investigator has exacerbated or contributed to the current headache pattern of the subject. Overuse is defined as an average of 10 days per month over the last 6 months.
14. has taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
15. is currently taking and plans to continue an oral steroid any time from screening through onset of menses that will be treated with study medication (at the discretion of the investigator)
16. has history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent.
17. has evidence or history of any gastrointestinal surgery or gastrointestinal (GI) ulceration or perforation in the past six months, gastrointestinal bleeding in the past year; or evidence or history of inflammatory bowel disease
18. is pregnant, actively trying to become pregnant, or breast feeding
19. has evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
20. has participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - Clinvest, Springfield, Missouri
  - University Internal Medicine Associates, Inc., Cincinnati, Ohio

REFERENCES:
- [Background] Martin VT, Behbehani M. Ovarian hormones and migraine headache: understanding mechanisms and pathogenesis--part 2. Headache. 2006 Mar;46(3):365-86. doi: 10.1111/j.1526-4610.2006.00370.x. PMID 16618254
- [Background] Martin VT, Wernke S, Mandell K, Ramadan N, Kao L, Bean J, Liu J, Zoma W, Rebar R. Symptoms of premenstrual syndrome and their association with migraine headache. Headache. 2006 Jan;46(1):125-37. doi: 10.1111/j.1526-4610.2006.00306.x. PMID 16412160
- [Background] Cady R, Dodick DW. Diagnosis and treatment of migraine. Mayo Clin Proc. 2002 Mar;77(3):255-61. doi: 10.4065/77.3.255. PMID 11888029
- [Background] Durham PL. Calcitonin gene-related peptide (CGRP) and migraine. Headache. 2006 Jun;46 Suppl 1(Suppl 1):S3-8. doi: 10.1111/j.1526-4610.2006.00483.x. PMID 16927957
- [Background] Nappi RE, Sances G, Brundu B, De Taddei S, Sommacal A, Ghiotto N, Polatti F, Nappi G. Estradiol supplementation modulates neuroendocrine response to M-chlorophenylpiperazine in menstrual status migrainosus triggered by oral contraception-free interval. Hum Reprod. 2005 Dec;20(12):3423-8. doi: 10.1093/humrep/dei260. Epub 2005 Aug 25. PMID 16123089
- [Background] Bellamy JL, Cady RK, Durham PL. Salivary levels of CGRP and VIP in rhinosinusitis and migraine patients. Headache. 2006 Jan;46(1):24-33. doi: 10.1111/j.1526-4610.2006.00294.x. PMID 16412148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects between the ages of 18 and 45 were recruited from two investigative sites. Subjects were enrolled from May 9,2011 through March 29, 2012. Last patient out June 5,2012.
Pre-assignment Details: Subjects were enrolled and randomized at Visit 1. There were no significant events between enrollment and assignment.
Groups:
- Placebo: Subjects randomized to Group B will be provided with 1 tablet of placebo to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Placebo : A placebo tablet matching Treximet for oral administration.
- Treximet: Subjects randomized to Group A will be provided with 1 tablet of Treximet to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Treximet : Tablet for oral administration contains sumatriptan 85mg / naproxen sodium 500mg.
Period: Overall Study
Arm/Group | Placebo | Treximet
Started | 20 | 21
Completed | 11 | 14
Not Completed | 9 | 7
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Subject withdrew due to personal issues. | 3 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treximet | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.35 (8.22) | 36.71 (6.50) | 35.56 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Migraine Recurrence
Description: Number of subjects either pain free or mild at 2 hours then pain level increases within 24 hours following treatment with Treximet versus (vs.) Placebo for 1 menstrual migraine.
  0-3 pain scale with 0=No Pain, 1=Mild, 2=Moderate,and 3=Severe.
Time Frame: From onset of a single menstrual migraine episode to 24 hours post menstrual migraine treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 11 | 14
participants | 0 | 2

2. Primary Outcome: Time to Pain Free
Description: Duration of 1 menstrual migraine from time of treatment at menstrual migraine headache onset until pain free in Treximet vs. Placebo arms.
  0-3 pain scale with 0=No Pain, 1=Mild, 2=Moderate, and 3=Severe.
Time Frame: From onset of 1 menstrual migraine headache until pain free.
Population: In Group B, one subject did not report when their headache resolve, therefore a duration for this subject could not be calculated.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
hours | 7.64 (4.06) | 3.90 (3.92)

3. Primary Outcome: Biomarkers Measured at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment
Description: Vasoactive Intestinal Peptide (VIP), Prostaglandin E2 (PGE2), Cortisol, Prostaglandin I2 (PGI2), Estradiol, and β-endorphin** levels collected at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Treximet vs. Placebo arms for 1 menstrual migraine headache * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure. Calcitonin Gene-Related Peptide (CGRP) and α-amylase both have their own outcome measure reported individually.
  **β-endorphin levels were not assayed due to limitations on saliva sample volumes.
Time Frame: From Baseline until 2 hours post treatment of 1 menstrual migraine headache
Population: In Group B, one subject's sample was unable to be analyzed by the laboratory, therefore Group B has one less subject in the placebo arm (N=10) for all biomarker data. Sample size for each arm may vary at each time point and/or biomarker based on laboratory results obtained due to sample collection errors.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
pg/mL
  VIP Baseline (n=10, 14) | 763.6 (341.01) | 1149.5 (532.07)
  VIP Migraine Onset (n=10, 13) | 1052.8 (490.57) | 1111.31 (560.39)
  VIP 2 Hours Post Treatment (n=9, 13) | 1130.44 (600.29) | 933.77 (643.38)
  PGE2 Baseline (n=10, 14) | 9.25 (7.97) | 12.65 (11.33)
  PGE2 Migraine Onset (n=10, 13) | 7.56 (2.61) | 13.02 (7.55)
  PGE2 2 Hours Post Treatment (n=9, 14) | 8.29 (4.43) | 7.99 (4.37)
  Cortisol Baseline (n=10, 13) | 1064.14 (970.57) | 1040.49 (1292.8)
  Cortisol Migraine Onset (n=8, 13) | 1084.85 (758.46) | 1209.34 (1795.19)
  Cortisol 2 Hours Post Treatment (n=8, 10) | 2011.45 (2259.76) | 418.48 (211.93)
  PGI2 Baseline (n=10, 14) | 109.51 (62.90) | 160.27 (100.22)
  PGI2 Migraine Onset (n=10, 13) | 108.23 (61.25) | 158.29 (76.74)
  PGI2 2 Hours Post Treatment (n=9, 14) | 97.58 (54.70) | 201.60 (115.16)
  Estradiol Baseline (n=10, 13) | 63.37 (42.24) | 62.61 (78.16)
  Estradiol Migraine Onset (n=9, 13) | 41.68 (30.43) | 43.93 (36.85)
  Estradiol 2 Hours Post Treatment (n=9,14) | 54.07 (36.45) | 41.66 (22.19)

4. Primary Outcome: CGRP Measured at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment
Description: CGRP levels collected at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Treximet vs. Placebo arms for 1 menstrual migraine headache
  * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
Time Frame: From Baseline until 2 hours post treatment for 1 menstrual migraine headache
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
pmol/mg
  CGRP Baseline (n=10, 14) | 18.55 (16.98) | 15.03 (11.73)
  CGRP Migraine Onset (n=10, 13) | 22.28 (14.45) | 27.82 (36.66)
  CGRP 2 Hours Post Treatment (n=9, 14) | 14.92 (11.96) | 21.38 (11.45)

5. Primary Outcome: α-Amylase Measured at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment
Description: α-Amylase levels collected at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Treximet vs. Placebo arm for 1 menstrual migraine headache
  * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
Time Frame: From Baseline until 2 hours post treatment for 1 menstrual migraine headache
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
U/L
  α-Amylase Baseline (n=10, 14) | 109280.50 (12499.73) | 99626.61 (7616.14)
  α-Amylase Migraine Onset (n=10, 13) | 100956.70 (13551.51) | 98853.32 (12958.58)
  α-Amylase 2 Hours Post Treatment (n=9, 14) | 102449.80 (4883.00) | 103594.90 (9335.72)

6. Secondary Outcome: Migraine Recurrence Responders vs Non-Responders
Description: Number of subjects either pain-free or mild at 2 hours then pain level increases within 24 hours following treatment in Treximet vs. Placebo arm for 1 menstrual migraine headache with Treximet vs. Placebo in responders* vs. non-responders.
  0-3 Pain Scale with 0=No Pain, 1=Mild, 2=Moderate, and 3=Severe
  *A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From the onset of 1 menstrual migraine until 24 hours post treatment.
Measure: Number; unit: participants
Groups:
- Treximet Responder: Subjects randomized to Group A will be provided with 1 tablet of Treximet to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Responders were defined as subjects who had a headache with a severity of 0=No Pain or 1=Mild Pain at two hours post treatment, and subjects could not have rescued with additional medication, and their headache could not have returned within 24 hours.
  Treximet : Tablet for oral administration contains sumatriptan 85mg / naproxen sodium 500mg.
- Treximet Non-Responder: Subjects randomized to Group A will be provided with 1 tablet of Treximet to be taken at onset of menstrual migraine headache pain.
  All subjects will be provided with 1 tablet of Treximet for treatment of persistent or recurring headache between 2 and 24 hours following treatment with study medication at headache onset.
  Non-Responders were defined as subjects who had a headache with a severity of 3=Severe Pain or 2=Moderate Pain at two hours post treatment, and/or subjects that rescued with additional medication, and/or their headache increased and/or returned within 24 hours.
  Treximet : Tablet for oral administration contains sumatriptan 85mg / naproxen sodium 500mg.
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 11 | 7 | 7
participants | 1 | 2 | 0

7. Secondary Outcome: Time to Pain-Free in Responders vs Non-Responders
Description: Duration of time from treatment at menstrual migraine headache onset until pain-free in Treximet vs. Placebo arms in responders* vs. non-responders for 1 menstrual migraine.
  0-3 Pain Scale, with 0=No Pain, 1=Mild, 2=Moderate, and 3=Severe.
  *A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From the onset of 1 menstrual migraine headache until pain-free.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
hours | 7.64 (4.06) | 3.13 (4.05) | 4.68 (3.93)

8. Secondary Outcome: Biomarkers Measured at Baseline, Menstrual Migraine Onset, and 2 Hours Post Treatment in Responders vs Non-Responders
Description: VIP, PGE2, Cortisol, PGI2, Estradiol, and β-endorphin** levels collected for 1 menstrual migraine headache at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Treximet vs. Placebo arms in responders vs. non-responders***.
  *This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same unit of measure. CGRP and α-amylase both have their own outcome measure reported individually.
  **β-endorphin levels were not assayed due to limitations on saliva sample volumes.
  ***A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline until 2 Hours post menstrual migraine treatment for 1 menstrual migraine headache.
Population: Sample size for each arm may vary at each time point and/or biomarker based on laboratory results obtained due to sample collection errors.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
pg/mL
  VIP Baseline (n=10,7,7) | 763.6 (341.01) | 1414.0 (618.96) | 885.0 (258.91)
  VIP Migraine Onset (n=10,7,6) | 1052.8 (490.57) | 1251.14 (580.38) | 948.17 (538.67)
  VIP 2 Hours Post Treatment (n=9,7,6,) | 1130.44 (600.29) | 1320.14 (657.68) | 414.0 (226.53)
  PGE2 Baseline (n=10,7,7) | 9.25 (7.97) | 14.29 (12.12) | 11.01 (11.12)
  PGE2 Migraine Onset (n=10,7,6) | 7.56 (2.61) | 14.13 (9.48) | 11.72 (5.02)
  PGE2 2 Hours Post Treatment (n=9,7,7) | 8.29 (4.43) | 6.83 (4.97) | 9.15 (3.69)
  Cortisol Baseline (n=10,6,7) | 1064.14 (970.57) | 790.77 (633.65) | 1254.53 (1700.66)
  Cortisol Migraine Onset (n=8,7,6) | 1084.5 (758.46) | 952.52 (864.35) | 1508.97 (2576.41)
  Cortisol 2 Hours Post Treatment (n=8,6,4) | 2011.45 (2259.76) | 482.32 (253.59) | 322.72 (84.78)
  PGI2 Baseline (n=10,7,7) | 109.51 (62.90) | 142.99 (65.71) | 177.54 (129.41)
  PGI2 Migraine Onset (n=10,7,6) | 108.23 (61.25) | 134.40 (71.0) | 186.17 (79.71)
  PGI2 2 Hours Post Treatment (n=9,7,7) | 97.58 (54.70) | 155.56 (63.48) | 247.63 (140.58)
  Estradiol Baseline (n=9,7,6) | 63.37 (42.24) | 49.60 (54.34) | 66.68 (98.50)
  Estradiol Migraine Onset (n=8,7,6) | 37.05 (31.67) | 44.89 (41.81) | 42.81 (34.04)
  Estradiol 2 Hours Post Treatment (n=8,7,7) | 54.07 (36.45) | 36.64 (23.20) | 46.68 (21.67)

9. Secondary Outcome: CGRP Measured at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post-Treatment in Responders vs Non-Responders
Description: CGRP levels collected for 1 menstrual migraine headache at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post-Treatment in Responders vs Non-Responders**.
  *This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
  **A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline until 2 Hours post menstrual migraine treatment for 1 menstrual migraine headache.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
pmol/mg
  CGRP Baseline (n=10,7,7) | 18.55 (16.98) | 12.27 (6.61) | 17.80 (15.39)
  CGRP Migraine Onset (n=10,7,6) | 22.28 (14.45) | 22.74 (11.94) | 33.76 (54.55)
  CGRP 2 Hours Post Treatment (n=9,7,7) | 14.92 (11.96) | 21.08 (8.02) | 21.67 (14.81)

10. Secondary Outcome: α-Amylase Measured at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Responders vs Non-Responders
Description: α-Amylase levels collected at Baseline, Menstrual Migraine Headache Onset, and 2 Hours Post Treatment in Responders vs Non-Responders*.
  *A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline until 2 hours post treatment of 1 menstrual migraine headache.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
U/L
  α-Amylase Baseline (n=10,7,7) | 109280.50 (12499.73) | 98002.68 (6613.71) | 101250.54 (8705.42)
  α-Amylase Migraine Onset (n=10,7,6) | 100956.7 (13551.51) | 103478.94 (10789.63) | 93456.77 (14086.68)
  α-Amylase 2 Hours Post Treatment (n=9,7,7) | 102449.88 (4883.0) | 103527.5 (12084.79) | 103662.4 (6540.98)

11. Primary Outcome: Biomarkers Measured at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free.
Description: VIP, PGE2, Cortisol, PGI2, Estradiol, and β-endorphin** levels collected at Menstrual Migraine Headache Onset, Migraine Headache Free and 24 Hours Migraine Headache Free in Treximet vs. Placebo arm for 1 menstrual migraine headache.
  * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure. CGRP and α-amylase both have their own outcome measure reported individually.
  **β-endorphin levels were not assayed due to limitations on saliva sample volumes.
Time Frame: From baseline to 24 hours post headache gone for 1 menstrual migraine headache.
Population: In Group B, one subject's sample was unable to be analyzed by the laboratory, therefore Group B has one less subject in the placebo arm (N=10) for all biomarker data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
pg/mL
  VIP Migraine Onset (n=10,7,6) | 1052.8 (490.57) | 1111.31 (560.39)
  VIP Migraine Headache Free (n=9,4,7) | 964.4 (711.43) | 949.7 (536.21)
  VIP 24 Hours Migraine Headache Free (n=10,7,6) | 1059.9 (564.42) | 1353.04 (629.56)
  PGE2 Migraine Onset (n=10,7,6) | 7.56 (2.61) | 13.02 (7.55)
  PGE2 Migraine Headache Free (n=10,4,6,) | 8.35 (6.52) | 9.27 (6.74)
  PGE2 24 Hours Migraine Headache Free (n=10,7,7) | 10.46 (11.43) | 13.04 (12.03)
  Cortisol Migraine Onset (n=8,7,6) | 1084.5 (7584.6) | 1209.34 (1795.19)
  Cortisol Migraine Headache Free (n=10,3,6) | 1490.92 (2232.7) | 1498.92 (1945.6)
  Cortisol 24 Hours Migraine Headache Free(n=10,6,6) | 1031.16 (1474.05) | 1271.4 (1606.11)
  PGI2 Migraine Onset (n=10,7,6) | 108.23 (61.25) | 158.29 (76.74)
  PGI2 Migraine Headache Free (n=10,4,6) | 115.63 (78.71) | 167.48 (94.28)
  PGI2 24 Hours Migraine Headache Free (n=10,7,7) | 97.69 (63.84) | 224.58 (160.51)
  Estradiol Migraine Onset (n=9,7,6) | 37.05 (31.67) | 43.93 (36.85)
  Estradiol Migraine Headache Free (n=9,4,5,) | 48.83 (48.82) | 39.92 (45.55)
  Estradiol 24 Hours Migraine Headache Free(n=6,7,5) | 21.34 (26.35) | 56.33 (53.49)

12. Primary Outcome: CGRP Measured at Menstrual Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free.
Description: CGRP levels collected at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Treximet vs. Placebo arm for 1 menstrual migraine headache.
  * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
Time Frame: From baseline to 24 hours post headache gone for 1 menstrual migraine headache
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
pmol/mg
  CGRP Migraine Onset (n=10,7,6) | 22.28 (14.45) | 28.82 (36.66)
  CGRP Migraine Headache Free (n=9,4,6) | 22.55 (30.87) | 32.26 (34.89)
  CGRP 24 Hours Migraine Headache Free (n=9,7,7) | 29.37 (26.76) | 32.15 (27.74)

13. Primary Outcome: α-Amylase Measured at Menstrual Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free.
Description: α-Amylase levels collected at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Treximet vs. Placebo arm for 1 menstrual migraine headache
  * This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
Time Frame: From baseline to 24 hours post headache gone for 1 menstrual migraine headache
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 10 | 14
U/L
  α-Amylase Migraine Onset (n=10,7,6) | 100956.70 (13551.51) | 98853.32 (12958.58)
  α-Amylase Migraine Headache Free (n=10,4,6) | 102908.61 (11522.83) | 101307.25 (8347.11)
  α-Amylase 24 Hours Migraine Headache Free(n=10,7,7 | 100354.00 (16608.96) | 102017.80 (8825.01)

14. Primary Outcome: Correlation of Mean Estrogen Levels in Saliva and Urine Estradiol at Mid Luteal and at Menstrual Migraine Headache Free.
Description: Correlation of mean estrogen levels in saliva and urine estradiol at mid luteal, menstrual migraine headache onset*, and at migraine headache free following treatment with Treximet vs. Placebo for 1 menstrual migraine headache
  *Urine estradiol levels were not collected at migraine onset, therefore; correlations could not be completed for that time point.
Time Frame: From mid luteal phase and for the duration of 1 menstrual migraine headache and until headache free
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet
Number analyzed (Participants) | 11 | 14
pg/mL
  Urine Pre-Cycle Day 1 (n=3, 6) | 2442.44 (545.38) | 3090.92 (2306.67)
  Urine Pre-Cycle Day 2 (n=6, 8) | 4333.92 (2982.35) | 2616.64 (2833.28)
  Urine Pre-Cycle Day 3 (n=8, 6) | 3582.92 (4121.17) | 5089.63 (5775.30)
  Urine Pre-Cycle Day 4 (n=9, 10) | 3232.10 (2941.52) | 3141.51 (2237.74)
  Urine Migraine Headache Free (n=11, 13 | 2398.55 (1872.88) | 2989.72 (3823.33)
  Saliva Pre-Cycle Day 1 (n=1, 4) | 41.75 (NA) — Only one subject's level was reportable for this single collection time point, therefore; mean and standard deviation could not be calculated with only one reported value. | 43.33 (23.19)
  Saliva Pre-Cycle Day 2 (n=2, 6) | 63.45 (57.60) | 41.87 (17.73)
  Saliva Pre-Cycle Day 3 (n=8, 10) | 46.47 (34.73) | 73.08 (58.17)
  Saliva Pre-Cycle Day 4 (n=6, 9) | 55.86 (50.17) | 41.72 (31.69)
  Saliva Migraine Headache Free (n=8, 6) | 54.93 (48.38) | 51.32 (45.64)

15. Secondary Outcome: Biomarkers Measured at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders
Description: VIP, PGE2, Cortisol, PGI2, Estradiol, and β-endorphin** levels collected for 1 menstrual migraine headache at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders***.
  *This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure. CGRP and α-amylase both have their own outcome measure reported individually.
  **β-endorphin levels were not assayed due to limitations on saliva sample volumes.
  ***A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment. A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline for the duration of 1 menstrual migraine headache, an estimated 7 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
pg/mL
  VIP Migraine Onset (n=10,7,6) | 105.28 (490.97) | 1251.14 (580.38) | 948.97 (538.67)
  VIP Migraine Headache Free (n=9,4,6) | 964.4 (711.43) | 1409.75 (567.81) | 643.0 (204.69)
  VIP 24 Hours Migraine Headache Free (n=10,7,5) | 1059.9 (564.42) | 1480.79 (624.74) | 1174.2 (660.26)
  PGE2 Migraine Onset (n=10,7,6) | 7.56 (2.61) | 14.13 (9.48) | 11.72 (5.02)
  PGE2 Migraine Headache Free (n=10,4,6) | 8.35 (6.52) | 7.87 (1.44) | 10.21 (8.82)
  PGE2 24 Hours Migraine Headache Free (n=10,7,7) | 10.46 (11.43) | 13.43 (14.38) | 12.65 (10.31)
  Cortisol Migraine Onset (n=8,7,6) | 1084.5 (758.46) | 952.52 (864.35) | 1508.97 (2576.41)
  Cortisol Migraine Headache Free (n=10,3,5) | 1490.92 (2232.7) | 592.35 (316.8) | 2042.87 (2363.89)
  Cortisol 24 Hours Migraine Headache Free(n=10,6,6) | 1031.16 (1474.05) | 863.09 (687.42) | 1621.38 (2110.87)
  PGI2 Migraine Onset (n=10,7,6) | 108.23 (61.25) | 134.40 (71.0) | 186.17 (79.71)
  PGI2 Migraine Headache Free (n=10,4,6) | 115.63 (78.71) | 154.16 (68.28) | 176.37 (113.87)
  PGI2 24 Hours Migraine Headache Free (n=10,7,7) | 97.69 (63.84) | 154.10 (71.61) | 295.07 (197.73)
  Estradiol Migraine Onset (n=9,7,6) | 37.75 (31.67) | 44.89 (41.81) | 42.81 (34.04)
  Estradiol Migraine Headache Free (n=9,5,4) | 48.83 (48.82) | 56.59 (67.39) | 26.58 (15.60)
  Estradiol 24 Hours Migraine Headache Free(n=6,7,6) | 21.34 (26.35) | 34.86 (46.64) | 81.38 (53.46)

16. Secondary Outcome: CGRP Measured at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders
Description: CGRP levels collected for 1 menstrual migraine headache at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders**.
  *This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
  **A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline to 24 hours post headache gone for 1 menstrual migraine.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pmol/mg
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
pmol/mg
  CGRP Migraine Onset (n=10,7,6) | 22.28 (14.45) | 22.74 (11.94) | 33.76 (54.55)
  CGRP Migraine Headache Free (n=9,4,6) | 22.55 (30.87) | 49.48 (49.68) | 20.78 (17.73)
  CGRP 24 Hours Migraine Headache Free (n=9,7,7) | 29.37 (26.76) | 28.43 (25.46) | 35.87 (31.41)

17. Secondary Outcome: α-Amylase Measured at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders
Description: α-Amylase levels collected for 1 menstrual migraine at Menstrual Migraine Headache Onset, Migraine Headache Free, and 24 Hours Migraine Headache Free in Responders vs Non-Responders**.
  *This endpoint was separated into 3 outcome measures as all biomarkers were not reported in the same units of measure.
  **A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From Baseline from 24 hours post migraine gone for 1 menstrual migraine.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
U/L
  α-amylase Migraine Onset (n=10,7,6) | 100956.7 (13551.51) | 103478.94 (10789.63) | 93456.77 (14086.08)
  α-amylase Migraine Headache Free (n=9,7,7) | 102908.61 (11522.83) | 98720.95 (13045.21) | 103031.44 (3793.21)
  α-amylase 24 Hours Migraine Headache Free(n=10,4,6 | 100354.3 (16608.96) | 102475.8 (9769.4) | 101559.9 (8532.96)

18. Secondary Outcome: Correlation of Mean Estrogen Levels in Saliva and Urine Estradiol at Mid-Luteal and at Menstrual Migraine Headache Free in Responders vs Non-Responders
Description: Correlation of mean estrogen levels in saliva and urine estradiol at mid-luteal, menstrual migraine headache onset* and at migraine headache free following treatment in responders vs. non-responders**.
  *Urine estradiol levels were not collected at migraine onset, therefore; correlations could not be completed for that time point.
  ***A responder is defined as those who at the time of two hours post treatment reported mild or no pain. Additionally, these subjects could not have taken a rescue medication or have a pain level increase within 24 hours post treatment.
  A non-responder is one that fails to meet the responder criteria.
Time Frame: From mid luteal phase and for the duration of 1 menstrual migraine until headache free.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Treximet Responder | Treximet Non-Responder
Number analyzed (Participants) | 10 | 7 | 7
pg/mL
  Urine Pre-Cycle Day 1 (n=3,2,4) | 2442.44 (545.38) | 1898.63 (92.07) | 3687.07 (2728.27)
  Urine Pre-Cycle Day 2 (n=6,3,5) | 4333.92 (2982.35) | 875.34 (377.69) | 3661.52 (3215.32)
  Urine Pre-Cycle Day 3 (n=8,2,5) | 3582.92 (4121.17) | 3739.44 (1536.97) | 5629.71 (6940.06)
  Urine Pre-Cycle Day 4 (n=9,5,5) | 3232.10 (2941.52) | 2016.99 (1295.30) | 4266.02 (2535.29)
  Urine Migraine Headache Free (n=10,7,7) | 2398.55 (1872.88) | 2542.09 (3152.52) | 3373.40 (4536.70)
  Saliva Pre-Cycle Day 1 (n=1,0,4) | 41.75 (NA) — Only one Subject's level was reported for this time point, therefore; mean and standard deviation could not be calculated. | NA (NA) — Unable to report for this group and time point as samples were not provided by any subjects in this group. Therefore, the mean and standard deviation could not be calculated. | 43.33 (23.19)
  Saliva Pre-Cycle Day 2 (n=2,2,4) | 63.45 (57.60) | 30.89 (7.16) | 47.36 (19.65)
  Saliva Pre-Cycle Day 3 (n=8,4,7) | 46.47 (34.73) | 81.05 (60.64) | 67.76 (61.65)
  Saliva Pre-Cycle Day 4 (n=8,5,4) | 55.86 (50.17) | 31.71 (26.78) | 54.22 (36.69)
  Saliva Migraine Headache Free (n=8,3,4) | 54.93 (48.38) | 75.45 (68.38) | 33.22 (5.48)

ADVERSE EVENTS:
Arm/Group | Placebo | Treximet
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 6/20 | 7/21
OTHER ADVERSE EVENTS (reported when occurring in more than 3.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Treximet (N=21)
Dull Stomach Ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left Side Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Feeling of Upper Body Heaviness (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (2) | 3 (4)
Drowsiness (General disorders) | 0 (0) | 1 (1)
Right Leg Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shakiness (Nervous system disorders) | 0 (0) | 1 (1)
Worsening Headache (Nervous system disorders) | 0 (0) | 1 (1)
Right Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Post bunionectomy
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Head Pressure (Nervous system disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flushing of Neck (Vascular disorders) | 1 (1) | 0 (0)
Arms Felt Warm (Vascular disorders) | 1 (1) | 0 (0)
Flushing of Face (Vascular disorders) | 1 (1) | 0 (0)
Jaw Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abnormal Alanine Aminotransferase (ALT) (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No